CLINICAL TRIAL: NCT06260111
Title: Laser Photobiomodulation to Prevent Oral Mucositis and Functional Impairment Among Adult Hematologic Cancer Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Photobiomodulation for Oral Mucositis and Functional Impairments During Hematopoietic Stem Cell Transplantation
Acronym: POMFITT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other); Clínica Dávila (Other)
Responsible Party: Principal Investigator, Cinara Sacomori, Ph.D., Principal Investigator, Universidad del Desarrollo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SA23I0021
Record Dates: First submitted 2024-01-26; First posted 2024-02-15 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Hematologic Cancer
Keywords: Low level laser therapy; Hematopoietic stem cell transplantation; Oral mucositis; Physical fitness; Physical therapy
MeSH Terms: conditions — Hematologic Neoplasms; Stomatitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The design of the study consists of a randomized, controlled trial with parallel groups (photobiomodulation + usual care versus a control group with only usual care), allocation ratio of 1:1.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor will be blinded only for the secondary outcomes. The person responsible for statistical analyses will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Experimental): Photobiomodulation and usual care (education, cryotherapy, and mouth hygiene).
  Interventions: Device: Photobiomodulation; Other: Usual care
- Control group (Other): Usual care (education, cryotherapy, and mouth hygiene).
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation will be used in sessions of approximately 5 to 10 minutes each. An InGaIP diode laser will be used with the following parameters: wavelength of 660 nm, output power of 40 mW, and an energy density of 4 J/cm2 measured at the end of the fiber optic with 0.04 cm2 of section area. The laser will be applied at 10 points in each oral region, with an exposure time of 4 s per point, using 0.16 J of energy per point.
  The protocol was based on previous studies.
  Other Names: Low level laser therapy
  Arms: Photobiomodulation group
Other: Usual care — Usual care for oral mucositis includes education, cryotherapy, and mouth hygiene.

SUMMARY:
The goal of this clinical trial is to test the efficacy of laser photobiomodulation in adult hematologic cancer patients undergoing hematopoietic stem cell transplantation (HSCT). The main questions it aims to answer are: • Is photobiomodulation with laser in the oral cavity, compared to standard care, effective in preventing oral mucositis and functional impairments in adult patients receiving HSCT? • What is the level of patient´s acceptability of photobiomodulation with laser in the oral cavity during HSCT? Participants once a day will receive photobiomodulation (diode laser device) in their oral cavity from the first day of transplantation conditioning until third day post-transplant. Researchers will compare with usual care to see if photobiomodulation helps preventing oral mucositis and functional impairment.

DETAILED DESCRIPTION:
Background: Oral mucositis is a highly prevalent condition in individuals treated for hematologic neoplasms, primarily during hematopoietic stem cell transplantation (HSCT). This condition delays the recovery process, increasing infections, interventions, and hospital stays. To date, there are few experimental trials evaluating the use of photobiomodulation with laser for the management of oral mucositis and reporting its effect on functional outcomes in patients with hematologic cancer undergoing HSCT.

Aim: To evaluate the effectiveness and social acceptability of using photobiomodulation in the oral cavity to prevent mucositis and functional impairments in adult patients undergoing HSCT.

Methods: Randomized controlled clinical trial with parallel groups (intervention group with photobiomodulation versus a control group), assessor and statistician blinded. Participants and setting: 30 patients with hematologic neoplasms aged 18 to 65 undergoing HSCT at the Oncology and Bone Marrow Transplant Unit of Clínica Dávila. Primary outcome measures: Oral mucositis will be assessed on a daily basis with the World Health Organization Scale. Functional capacity will be evaluated with a 2-minute static walking test; handgrip strength using digital Jamar® dynamometry; lower limb strength with 30s Sits-and-Stand test; and quality of life using the Functional Assessment of Cancer Therapy Bone Marrow Transplant questionnaire. Acceptability will be assessed by recording treatment adherence and a Visual Analog Scale. Evaluations will be performed at two time points: on admission to the transplant unit before the start of the conditioning regimen and on the day of hospital discharge. Intervention: Photobiomodulation will be delivered from the first day of conditioning until day 3 post-transplant. A diode laser device with a wavelength of 660 nm, an output power of 40 mW, and an energy density of 4 J/cm2 measured at the end of the optical fiber with 0.04 cm2 of sectional area will be used. The investigators expect that photobiomodulation prevents oral mucositis and enhance functional capacity, muscle strength, nutritional status, and quality of life in patients with hematologic cancer undergoing bone marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age with hematological neoplasms who require medical indication of an HSCT according to the Transplant Committee at Clinica Dávila
* With sufficient understanding of Spanish.

Exclusion Criteria:

* Observed cognitive deficit
* Patients who do not meet the criteria of clinical stability, progression of the disease, and that do not fulfill requirement of the National Hematopoietic Stem Cell Transplantation Program.
* Participants with an oral infection from any type of Candida prior to HSCT.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Oral Mucositis | From the first day up to the 20th after stem cell transplantation (or up to the day of hospital discharge if prior to day 20)
  It refers to the maximal degree of oral mucositis developed after stem cell transplantation. It will be recorded daily from the first day after stem cell transplantation up to the day 20 after transplantation). The World Health Organization (WHO) oral mucositis scale will be used. Scores range from 0 (no mucositis), 1 (pain/erythema), 2 (erythema, ulcers; can eat solid foods), 3 (ulceration, requiring only a liquid diet), to 4 (oral feeding is not possible). The higher the grade, the worse the mucositis.
Level of Pain | From the first day up to the 20th day after stem cell transplantation (or up to the day of hospital discharge if prior to day 20)
  It refers to the perceived level of pain related to oral mucositis from a numeric scale (0 to 10), where 0 means "no pain" and 10 "the worse possible pain". Higher scores means more pain.

SECONDARY OUTCOMES:
Handgrip strength | Through study completion on the day of hospital discharge, an average of 1 month
  It is the maximal isometric strength of the handgrip that will be measured in KgF with Hydraulic Hand Dynamometer (Jamar Digital Plus®).
Exercise tolerance | Through study completion on the day of hospital discharge, an average of 1 month
  The exercise capacity of an individual as measured by endurance (maximal exercise duration and/or maximal attained work load) during an EXERCISE TEST. It will be assessed with the 2-Minute Walking Test is a functional test that assesses an individual's aerobic capacity and is used as a performance measure.
Physical fitness | Through study completion on the day of hospital discharge, an average of 1 month
  It is the ability to carry out daily tasks and perform physical activities in a highly functional state, often as a result of physical conditioning. Physical fitness will be evaluated with the 30-Second Sit and Stand (SST30') assesses the ability to rise from a chair and sit back down, as well as the strength and functionality of the lower limbs.
Health related quality of life | Through study completion on the day of hospital discharge, an average of 1 month
  Health related quality of life is a generic concept reflecting concern with the modification and enhancement of life attributes, e.g., physical, political, moral, social environment as well as health and disease. Quality of life will be assessed using the validated and widely used instrument in the oncology population undergoing hematopoietic stem cell transplantation, the Functional Assessment of Cancer Therapy-Bone Marrow Transplant questionnaire.
Length of hospital stay | Through study completion on the day of hospital discharge, an average of 1 month
  Number of hospitalization days/bed days from the day of admission to medical discharge
Use of opioids | Through study completion on the day of hospital discharge, an average of 1 month
  The number of days that the patient required analgesic medication (opioids) and receives it to alleviate oral mucositis pain from the onset of oral mucositis according to World Health Organization criteria until medical discharge.
Body mass index | Through study completion on the day of hospital discharge, an average of 1 month
  The body mass index is a person's weight in kilograms divided by the square of height in meters. It will be obtained from the patient's clinical file. Higher values mean malnutrition due to body weight excess and lower values mean malnutrition due to underweight. It will be classified according to World Health Organization: underweight (<18.5), normal weight (18,5 to 24.9), overweight (25 to 29.9) and obesity (>30).
Nutritional status | Through study completion on the day of hospital discharge, an average of 1 month
  Nutritional status has been defined as an individual's health condition as it is influenced by the intake and utilization of nutrients. The evaluation of the nutritional status will be through the Subjective Global Evaluation. This scale classifies patients in: well nourished, mildly/moderately malnourished, or severely malnourished.
Daily calorie intake | Through study completion on the day of hospital discharge, an average of 1 month
  It correspond to the mean of daily calorie intake (kcal/day) of the patient. It will be obtained from the hospital record. Higher values mean higher calorie intake.
Arm circumference | Through study completion on the day of hospital discharge, an average of 1 month
  It is the circumference of the arm (cm) that will be measured in the mean point between the distance of olecranon and acromion with relaxed arm and elbow flexed at 90 degrees.
Triceps skinfold | Through study completion on the day of hospital discharge, an average of 1 month
  Corresponds to the thickness of the triceps region (mm). It will be assessed with a skinfold caliper. Higher values indicate more body fat.
Acceptability | Through study completion on the day of hospital discharge, an average of 1 month
  To estimate patient´s acceptability, a visual analogue scale from 0 to 10 will be used only with intervention group, where 0 refers to no acceptability, 5 to a moderate level of acceptability and 10 to an optimal level of acceptability. Furthermore, the register of adherence to the PBM sessions will serve as an indicator of this acceptability, since the professional who performs the intervention will consult the patient every day regarding their willingness to receive PBM and will note on the record sheet.
Number of days from transplant to engraftment | Through study completion on the day of hospital discharge, an average of 1 month
  It to refers to how long, in days, did it take to engrafment of the hematopoyetic stem cell transplant. Engraftment is the process by which hematopoietic stem cells (HSC) make their way (homing) to free bone marrow (BM) niches where they can find optimal conditions to survive and proliferate.

CONTACTS AND LOCATIONS:
Overall Officials: Cinara Sacomori, Ph.D., Principal Investigator — Universidad del Desarrollo; Paulina A Araya-Castro, Ph.D., Study Chair — Universidad del Desarrollo
Locations (1):
- Clinica Dávila, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be requested to the researchers by e-mail, in case of relevant justification. All data shared with other researchers will be anonymous.
Supporting Information: Study Protocol, SAP
Time Frame: Data of study protocol will be available from the completion of the study up to 10 years after.
Access Criteria: Regulatory institutions such as Ethical Committee Board and Funding Audits will have full access to IPD if they require so.

REFERENCES:
- [Background] Ferreira B, da Motta Silveira FM, de Orange FA. Low-level laser therapy prevents severe oral mucositis in patients submitted to hematopoietic stem cell transplantation: a randomized clinical trial. Support Care Cancer. 2016 Mar;24(3):1035-42. doi: 10.1007/s00520-015-2881-8. Epub 2015 Aug 7. PMID 26248655
- [Background] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Background] Robijns J, Nair RG, Lodewijckx J, Arany P, Barasch A, Bjordal JM, Bossi P, Chilles A, Corby PM, Epstein JB, Elad S, Fekrazad R, Fregnani ER, Genot MT, Ibarra AMC, Hamblin MR, Heiskanen V, Hu K, Klastersky J, Lalla R, Latifian S, Maiya A, Mebis J, Migliorati CA, Milstein DMJ, Murphy B, Raber-Durlacher JE, Roseboom HJ, Sonis S, Treister N, Zadik Y, Bensadoun RJ. Photobiomodulation therapy in management of cancer therapy-induced side effects: WALT position paper 2022. Front Oncol. 2022 Aug 30;12:927685. doi: 10.3389/fonc.2022.927685. eCollection 2022. PMID 36110957
- [Background] Tribolet P, Kaegi-Braun N, Gressies C, Baumgartner A, Wagner KH, Stanga Z, Schuetz P. Handgrip Strength Values Depend on Tumor Entity and Predict 180-Day Mortality in Malnourished Cancer Patients. Nutrients. 2022 May 23;14(10):2173. doi: 10.3390/nu14102173. PMID 35631314
- [Background] Bohannon RW, Crouch RH. Two-Minute Step Test of Exercise Capacity: Systematic Review of Procedures, Performance, and Clinimetric Properties. J Geriatr Phys Ther. 2019 Apr/Jun;42(2):105-112. doi: 10.1519/JPT.0000000000000164. PMID 29210933
- [Background] McQuellon RP, Russell GB, Cella DF, Craven BL, Brady M, Bonomi A, Hurd DD. Quality of life measurement in bone marrow transplantation: development of the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) scale. Bone Marrow Transplant. 1997 Feb;19(4):357-68. doi: 10.1038/sj.bmt.1700672. PMID 9051246
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Derived] Lopez-Espinoza T, Sacomori C, Araya-Castro P, Quintiliano-Scarpelli D, Roldan P, Pena-Espinoza M, de Rezende LF, Lopez-Vidal H. Photobiomodulation therapy to prevent oral mucositis and functional impairment in adult patients with haematological cancer undergoing haematopoietic stem cell transplantation: randomised trial protocol. BMJ Open. 2024 Oct 26;14(10):e088073. doi: 10.1136/bmjopen-2024-088073. PMID 39461860
- See also: Definition of outcomes — https://www.ncbi.nlm.nih.gov/mesh/